CLINICAL TRIAL: NCT04032899
Title: Multicenter, Randomized, Double-blind, Controlled Parallel Nutritional Intervention Study to Evaluate the Effect of Consumption During Pregnancy and the Lactation Period of Lactobacillus Fermentum CECT5716 on the Incidence of Mastitis
Brief Title: Effect of Probiotics Consumed During Pregnancy on the Incidence of Mastitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P045
Record Dates: First submitted 2019-05-27; First posted 2019-07-25 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Mastitis; Breast Milk; Lactation; Women's Health; Infant Health
Keywords: Probiotics; Gestation; Lactation; Mastitis
MeSH Terms: conditions — Mastitis; Breast Feeding | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L. fermentum CECT5716 3x109 ufc (Experimental): Volunteers will take 1 capsule per day with L. fermentum CECT5716 3x109 cfu mixed with maltodextrin from week 28-32 of gestation up to 16 weeks after delivery.
  Interventions: Dietary Supplement: Lactobacillus fermentum CECT5716
- Maltodextrin (Placebo Comparator): Volunteers will take 1 capsule per day with maltodextrin from week 28-32 of gestation up to 16 weeks after delivery.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Lactobacillus fermentum CECT5716 — Each participant will consume 1 capsule per day in one of the main meals without any restriction in the diet or in their life habits.
  Arms: L. fermentum CECT5716 3x109 ufc
Dietary Supplement: Maltodextrin — Each participant will consume 1 capsule per day in one of the main meals without any restriction in the diet or in their life habits.
  Arms: Maltodextrin

SUMMARY:
The aim of the present study is to evaluate the effect of consumption during pregnancy and the lactation period of the probiotic L. fermentum CECT5716 on the incidence of mastitis.

Bacterial load and immunological parameters in breast milk, parameters related to breastfeeding as well as health parameters of the mother and baby will also be evaluated.

DETAILED DESCRIPTION:
Pregnancy and lactation are important moments for the child that will determine their development and future health. One of the key processes is when the microbiota is established in the baby. Contamination during delivery with the mother's vaginal flora, as well as bacteria from the microbiota of breast milk, are important sources for intestinal colonization. However, the mother's microbiota can suffer alterations that affect the health of the mother and can also have an effect on the baby.

Mastitis is a condition of the mammary gland that can affect between 3-30% of women during the period of lactation and is the first cause of abandonment of it. It is associated with a dysbiosis with the proliferation of microorganisms in milk such as Staphylococcus and Streptococcus.

Previous studies carried out with the strain L. fermentum CECT5716 have demonstrated a powerful regulating activity of the microbiota of breast milk that translates into a preventive and curative effect on mastitis. The highest incidence of mastitis occurs during the first weeks after delivery, so the investigator's working hypothesis is that the modulation of the maternal microbiota before delivery would improve the effectiveness of the probiotic strain consumption.

ELIGIBILITY:
Inclusion Criteria:

* Normal development of pregnancy
* Single fetus pregnancy
* Be in week 28-32 of pregnancy
* Intention to breastfeed the child for 16 weeks

Exclusion Criteria:

* Having a breast disease that hinders or prevents breastfeeding
* Have been taking probiotic supplements 2 weeks before starting the study
* Have a low expectation of adherence to the study protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 480 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of mastitis | 4 months
  Total events during breastfeeding period /total number of participants

SECONDARY OUTCOMES:
Microbiota of breast milk | 4 months
  Load of Staphylococcus, S. aureus, S. epidermidis, Streptococcus, Lactobacillus and L. fermentum CECT5716 in breast milk

OTHER OUTCOMES:
Recurrence of mastitis | 4 months
  Reappearance of mastitis symptoms
Breast pain questionnaire | 4 months
  Mcgill Pain Questionnaire, validated for Spain. The Questionnaire has four dimensions or scales of measures of intensity: Sensory Intensity Value, Affective Intensity Value, Current Intensity Value, and Evaluative Intensity Value. The scales of the Questionnaire were calculated as the sum of their items. Those items were re-corded as 1 if the participant described the pain or as 0 if the participant did not report that type of pain. Thus, the sensory intensity scale can range from 0 to 33, as the full scale is formed by 33 items. The Affective scale varies from 0 to 19, and the scales of Current Intensity and Evaluative Intensity can range from 0 to 6 and 5, respectively
Time of Breastfeeding | 4 months
  Date of initiation and cessation of breastfeeding
Percentage of infants breastfeed | 4 months
  Percentage of infants who receive exclusive breastfeeding
Measurement of biomarkers of inflammation in breast milk | 4 months
  Concentration of IL-1b, IL-6, IL-8, IL-17, TNF-α in breast milk
Immunoglobulins in breast milk | 4 months
  Concentration of IgA, IgG1, IgG2, IgG3, IgG4 and IgM in breast milk
Minerals in breast milk | 4 months
  Concentration of calcium (μg/L), magnesium (μg/L) and potassium (μg/L) in breast milk
Baby feces microbiota | 4 months
  Presence of Escherichia coli, Clostridium, Bacteroides, Bifidobacteria, Lactobacillus and L. fermentum CECT5716 in baby feces
Data on childbirth | 4 months
  Incidence of cesareans and incidence of antibiotic use during delivery.
Baby's anthropometric measures | 16 weeks
  Anthropometric measures of the baby (weight in kg, height in cm and BMI in kg/m2) at birth, 4 weeks, 8 weeks and 16 weeks.
Data about the intestinal health of the baby | 4 months
  Data about stool frequency, colour and consistency of the feces and gasses
Data about sleep parameters of the baby | 4 months
  Hours of night sleeping per day and hours of total sleeping during the day

CONTACTS AND LOCATIONS:
Overall Officials: Nicolás Mendoza, MD, PhD, Principal Investigator — Professor of Gynecology at the Faculty of Medicine of the University of Granada
Locations (3):
- Spain (3):
  - Hospital Costa del Sol, Marbella, Andalusia
  - Hospital Campus de la Salud, Granada, Grabada
  - Hospital Virgen de las Nieves, Granada, Granada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crepinsek MA, Taylor EA, Michener K, Stewart F. Interventions for preventing mastitis after childbirth. Cochrane Database Syst Rev. 2020 Sep 29;9(9):CD007239. doi: 10.1002/14651858.CD007239.pub4. PMID 32987448